CLINICAL TRIAL: NCT06074562
Title: A Phase 2, Randomized, Double-Blind, Placebo Controlled, Dose-Ranging Study to Evaluate LY3556050 in Adult Participants With Diabetic Peripheral Neuropathic Pain
Brief Title: A Study of LY3556050 in Adult Participants With Diabetic Peripheral Neuropathic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18509; J2P-MC-LXBD (Other: Eli Lilly and Company); 2023-506127-29-00 (Other: EU Trial Number)
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Diabetic Peripheral Neuropathy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LY3556050 Dose 1 (Experimental): Participants will receive LY3556050 orally.
  Interventions: Drug: LY3556050
- LY3556050 Dose 2 (Experimental): Participants will receive LY3556050 orally.
  Interventions: Drug: LY3556050
- LY3556050 Dose 3 (Experimental): Participants will receive LY3556050 orally.
  Interventions: Drug: LY3556050
- Placebo (Placebo Comparator): Participants will receive placebo orally.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3556050 — Administered orally.
  Arms: LY3556050 Dose 1; LY3556050 Dose 2; LY3556050 Dose 3
Drug: Placebo — Administered orally.
  Arms: Placebo

SUMMARY:
The main purpose of this study is to determine the safety and efficacy of LY3556050 versus placebo in participants with diabetic peripheral neuropathic pain (DPNP). The study will lasts approximately 24 weeks, across 3 study periods.

ELIGIBILITY:
Inclusion Criteria:

* Have a history and current diagnosis of Type 1 Diabetes (T1D) or Type 2 Diabetes (T2D) diagnosed for at least 6 months prior to screening.
* Have a stable glycemic control on stable diabetes treatment regimen for at least 90 days prior to day 1 with a hemoglobin A1c (HbA1c) ≤10 for T1D and HbA1c ≤11 for participants with T2D at time of screening.
* Have a history of daily peripheral neuropathic pain for at least 12 weeks based on participant report or medical history.
* Have a visual analog scale (VAS) pain value ≥40 and <95 during screening.
* Have presence of diabetic peripheral neuropathy of symmetrical nature and in lower extremities for ≥6 months and diagnosed by a score of Part B ≥3 on Michigan Neuropathy Screening Instrument
* Are willing to maintain a consistent regimen of any ongoing nonpharmacologic pain-relieving therapies (for example, physical therapy) and will not start any new nonpharmacologic pain-relieving therapies during study participation.
* Are willing to discontinue all medications taken for chronic pain conditions, except allowed concomitant pain medication permitted per protocol, for the duration of the study

  * Have a body mass index ≤45 kilogram/square meter (kg/m²) (inclusive).
  * Are men, or women able to abide by reproductive and contraceptive requirements.

Exclusion Criteria:

* History of other potentially causative and/or confounding sources of pain that may impair self-assessment of pain due to DPNP.
* Have had a procedure within the past 6 months intended to produce permanent sensory loss in the target area of interest (for example, ablation techniques.
* Have had cancer within 2 years of baseline, except for cutaneous basal cell or squamous cell carcinoma resolved by excision.
* Are, in the judgment of the investigator, actively suicidal and therefore deemed to be at significant risk for suicide.
* Have in the judgement of the investigator, an acute, serious, or unstable medical condition or a history or presence of any other medical illness that would preclude study participation.
* Have a positive HIV test result at screening.
* Have a surgery planned during the study for any reason.
* Have a substance use disorder as defined by the Diagnostic and Statistical Manual of Mental Disorders (5th edition; DSM-5; American Psychiatric Association)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2023-10-05 (Actual); Primary Completion 2025-06-11 (Actual); Study Completion 2025-06-11 (Actual)

PRIMARY OUTCOMES:
Mean Change from Baseline for Average Pain Intensity Numeric Rating Scale (API-NRS) | Baseline, Week 12

SECONDARY OUTCOMES:
Mean Change from Baseline for Worst Pain Intensity Numeric Rating Scale (WPI-NRS) | Baseline, Week 12
Mean Change from Baseline for Patient Reported Outcomes Measurement Information System (PROMIS) Pain Interference Short Form (SF)8a | Baseline, Week 12
Mean Change from Baseline for Pain Interference with Sleep | Baseline, Week 12
Mean Change from Baseline for PROMIS Physical Functioning Short Form (SF)10a | Baseline, Week 12
Mean Change from Baseline for PROMIS Sleep Disturbance (SD)8b | Baseline, Week 12
Mean Change from Baseline for Patient's Global Impression of Illness (PGI) Severity as Measured by PGI-Severity | Baseline, Week 12
Mean Change from Baseline for Patient's Global Impression of Illness Status as Measured by PGI-Status | Baseline, Week 12
Mean Change from Baseline for Patient's Global Impression of Change as Measured by PGI-Change | Baseline, Week 12
Mean Change from Baseline for Neuropathy Total Symptom Score-6 (NTSS-6) | Baseline, Week 12
Summary of Frequency, Timing and Amount of Rescue Medication Used During the Treatment Period | Baseline to Week 12
Pharmacokinetics (PK): Plasma Concentration of LY3556050 | Baseline to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (70):
- United States (34):
  - The Institute for Liver Health II dba Arizona Clinical Trials - Mesa, Chandler, Arizona
  - Headlands Research - Scottsdale, Scottsdale, Arizona
  - Orange Grove Family Practice, Tucson, Arizona
  - Preferred Research Partners, Little Rock, Arkansas
  - Hope Clinical Research, Inc., Canoga Park, California
  - Valley Clinical Trials, Inc., Northridge, California
  - Northern California Research - Sacramento, Sacramento, California
  - CMR of Greater New Haven, LLC, Hamden, Connecticut
  - Suncoast Research Group, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - Northwestern University, Chicago, Illinois
  - Alliance for Multispecialty Research, LLC, Wichita, Kansas
  - Alliance for Multispecialty Research, LLC, Lexington, Kentucky
  - Care Access - Lake Charles, Lake Charles, Louisiana
  - MedVadis Research Corporation, Waltham, Massachusetts
  - SKY Integrative Medical Center/SKYCRNG, Ridgeland, Mississippi
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Alliance for Multispecialty Research, LLC, Kansas City, Missouri
  - Clinvest Research LLC, Springfield, Missouri
  - Las Vegas Medical Research, Las Vegas, Nevada
  - UniMed Center, East Brunswick, New Jersey
  - North Suffolk Neurology, Port Jefferson Station, New York
  - Lucas Research - Hickory, Hickory, North Carolina
  - Lucas Research, Inc, Morehead City, North Carolina
  - Velocity Clinical Research, Medford, Medford, Oregon
  - Tristar Clinical Investigations, Philadelphia, Pennsylvania
  - Suburban Research Associates, West Chester, Pennsylvania
  - New Phase Research and Development, Knoxville, Tennessee
  - FutureSearch Trials of Neurology, Austin, Texas
  - Juno Research, Houston, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - Velocity Clinical Research, Salt Lake City, West Jordan, Utah
  - Northwest Clinical Research Center, Bellevue, Washington
  - Rainier Clinical Research Center, Renton, Washington
- Czechia (7):
  - EDUMED - Broumov, Broumov, Královéhradecký kraj
  - Diabet2 s.r.o., diabetologicka a interni ambulance, Prague, Praha 1
  - Neurologická Ambulance - Forbeli, Prague, Praha 6
  - DiaVize s.r.o., Prague, Praha, Hlavní Mešto
  - FLEDIP - Na dlouhem lanu, Prague, Praha, Hlavní Mešto
  - Vestra Clinics, European Union, Rychnov Nad Kněžnou
  - Agentura Science Pro, Olomouc
- Japan (13):
  - Matsuyama Shimin Hospital, Matsuyama, Ehime
  - Kikuchi Naika Clinic, Maebashi, Gunma
  - Kure Medical Center, Kure, Hiroshima
  - Japanese Red Cross Asahikawa Hospital, Asahikawa, Hokkaido
  - Yokohama Minoru Clinic, Yokohama, Kanagawa
  - Medical Corporation Heishinkai OCROM Clinic, Suita-shi, Osaka
  - Sugiura Internal Medicine Clinic, Sokashi, Saitama
  - Suruga Clinic, Shizuoka, Shizuoka
  - Medical Corporation Sato Medical clinic, Ootaku, Tokyo
  - Heishinkai Medical Group ToCROM Clinic, Shinjuku-ku, Tokyo
  - Kunisaki Makoto Clinic, Fukuoka
  - Minamiosaka Hospital, Osaka
  - Plumeria DM Clinic, Shizuoka
- Poland (11):
  - Nzoz Neuro-Kard Ilkowski i Partnerzy SPL, Poznan, Greater Poland Voivodeship
  - MICS Centrum Medyczne Torun, Torun, Kuyavian-Pomeranian Voivodeship
  - Medyczne Centrum Diabetologiczno Endokrynologiczno Metaboliczne DIAB-ENDO-MET, Krakow, Lesser Poland Voivodeship
  - Centrum Badań Klinicznych Piotr Napora lekarze sp.p., Wroclaw, Lower Silesian Voivodeship
  - MICS Centrum Medyczne Warszawa, Warsaw, Masovian Voivodeship
  - Samodzielny Publiczny Zespol Opieki Zdrowotnej w Wyszkow, Wyszków, Masovian Voivodeship
  - Zdrowie Osteo-Medic, Biaystok, Podlaskie Voivodeship
  - Centrum Medyczne Pratia Katowice, Katowice, Silesian Voivodeship
  - Pro Familia Altera, Katowice, Silesian Voivodeship
  - NZOZ Przychodnia Specjalistyczna Andrzej Wittek, Henryk Rudzki, Ruda Śląska, Silesian Voivodeship
  - Centrum Terapii Wspolczesnej J. M. Jasnorzewska Spolka Komandytowo-Akcyjna, Lodz, Łódź Voivodeship
- South Korea (5):
  - Sejong General Hospital, Sosa-gu, Kyǒnggi-do
  - Nowon Eulji Medical Center, Eulji University, Seoul, Seoul-teukbyeolsi [Seoul]
  - Konkuk University Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - Samsung Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - Eulji University Hospital, Daejeon, Taejǒn-Kwangyǒkshi

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: A Study of LY3556050 in Adult Participants With Diabetic Peripheral Neuropathic Pain — https://trials.lilly.com/en-US/trial/427360